CLINICAL TRIAL: NCT07106112
Title: A Randomized Trial Comparing Carbon Suspension (Black Eye) and Metallic Markers (TWIRL ULTRACOR) for Localization of Metastatic Axillary Lymph Nodes Prior to Neoadjuvant Systemic Therapy in Breast Cancer Patients.
Brief Title: Carbon Suspension vs. Metallic Marker for Axillary Lymph Node Marking in Breast Cancer After Neoadjuvant Therapy
Acronym: COMET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Alina Olchonova, Principal Investigator, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 05/45
Record Dates: First submitted 2025-07-24; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Carbon suspension; Axillary lymph node marking; Neoadjuvant therapy; Targeted axillary dissection; Metallic marker
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections; Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbon Suspension (Black Eye) Marking (Experimental)
  Interventions: Procedure: Ultrasound-guided carbon suspension (Black Eye) injection
- Metallic Marker (TWIRL ULTRACOR) Placement (Active Comparator)
  Interventions: Procedure: Ultrasound-guided metallic marker (TWIRL ULTRACOR) placement

INTERVENTIONS:
Procedure: Ultrasound-guided carbon suspension (Black Eye) injection — Under ultrasound guidance, 0.5 mL of sterile carbon particle suspension (Black Eye) is injected into the capsule of the metastatic axillary lymph node(s).
  Technique: Performed using a high-frequency linear ultrasound probe (e.g., 12 MHz) and a 22G needle.
  Target: Up to 3 pathologically confirmed metastatic lymph nodes. Timing: Performed before initiation of neoadjuvant systemic therapy (NST).
  Rationale:
  Carbon suspension provides long-term visual localization due to its black staining properties.
  Inert and biocompatible, with minimal risk of allergic reactions. Patients proceed to standard NST based on tumor subtype (chemotherapy, targeted therapy, or endocrine therapy).
  Post-NST imaging (ultrasound, CT, or PET-CT) to assess treatment response.
  Surgical Intervention:
  Targeted axillary dissection (TAD) with removal of marked nodes + sentinel lymph node biopsy (SLNB) using fluorescent dye.
  Intraoperative frozen section analysis (hematoxylin & eosin staining) of excised nodes.
  Arms: Carbon Suspension (Black Eye) Marking
Procedure: Ultrasound-guided metallic marker (TWIRL ULTRACOR) placement — A 4-mm nitinol (nickel-titanium alloy) marker (TWIRL ULTRACOR) is deployed into the metastatic lymph node(s) under ultrasound guidance.
  Technique: Uses a specialized introducer kit for precise placement. Target: Up to 3 pathologically confirmed metastatic lymph nodes. Timing: Performed before initiation of NST.
  Rationale:
  Nitinol markers are radiopaque, MRI-compatible, and resistant to migration. Standard method for tumor localization in breast cancer.
  Post-Marking Protocol:
  Identical NST and imaging follow-up as Group 1.
  Surgical Intervention:
  TAD with marker localization (palpation/imaging-guided excision) + SLNB. Intraoperative frozen section analysis.
  Arms: Metallic Marker (TWIRL ULTRACOR) Placement

SUMMARY:
This single-center, randomized study aims to compare the intraoperative detection rates of axillary lymph nodes marked with carbon suspension versus metallic markers in breast cancer patients (T1-3N1M0) before neoadjuvant therapy. Primary endpoint: frequency of marked lymph node identification during surgery. Secondary endpoints: time from marking to surgery and quality of life (EORTC QLQ-BR23).

DETAILED DESCRIPTION:
Interventions:

Group 1: Ultrasound-guided injection of 0.5 mL carbon suspension (Black Eye). Group 2: Ultrasound-guided placement of a metallic marker (TWIRL ULTRACOR). Follow-up: 6 months post-surgery. Design: Randomized 1:1, non-inferiority trial.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years.
* Morphologically confirmed breast cancer (T1-3N1M0).
* ECOG 0-1.
* Indication for neoadjuvant therapy.
* Signed informed consent.

Exclusion Criteria:

* No lymph node regression post-neoadjuvant therapy (persistent N1).
* Distant metastasis progression.
* Severe comorbidities (NYHA III-IV, COPD GOLD D, Child-Pugh C).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative detection rate of marked lymph nodes (%) | Assessed intraoperatively (day of surgery).
  The proportion of successfully identified and excised marked lymph nodes during surgery, confirmed by visual (carbon suspension) or imaging/metallic detection (metallic marker)

SECONDARY OUTCOMES:
Time from Marking to Surgery (Days) | From the date of marking procedure (Day 0) to the date of surgery (up to 12 weeks post-marking)
  Measures the duration (in days) between the lymph node marking procedure (carbon suspension or metallic seed placement) and the subsequent surgical intervention (targeted axillary dissection). This assesses the clinical feasibility and logistical timeline between marking and definitive treatment
Quality of Life (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Breast Cancer Module [EORTC QLQ-BR23] Scores | 1. Baseline (pre-marking), 2. Post-neoadjuvant therapy (pre-surgery) 3. 1-month postoperatively.
  Patient-reported outcomes assessed using the validated 23-item EORTC QLQ-BR23 questionnaire, which measures:
  Functional scales (Body Image, Sexual Functioning, Sexual Enjoyment, Future Perspective; higher scores = better outcomes), Symptom scales (Systemic Therapy Side Effects, Breast Symptoms, Arm Symptoms, Upset by Hair Loss; higher scores = worse outcomes).
  All items are scored 1-4 (raw scores) and transformed to a 0-100 scale. For functional scales, 100 represents optimal functioning; for symptom scales, 100 represents maximal symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Alina A Olchonova, Physician, Principal Investigator — Saint Petersburg State University, Russia
Locations (1):
- St. Petersburg State University, Saint Petersburg, Russia